CLINICAL TRIAL: NCT01846338
Title: The Effect of「GTT-EGCG」on Acne Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Chung-Hua Hsu, Associated Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCHIRB1010505
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Acne Lesion Counts
Keywords: acne, EGCG, green tea
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- green tea extract EGCG (Experimental): experimental: green tea extract EGCG, 500mg , tid, 4 weeks
  Interventions: Dietary Supplement: green tea extract EGCG
- cellulose (Placebo Comparator): Placebo Comparator: cellulose, 500 mg tid, 4 weeks
  Interventions: Dietary Supplement: green tea extract EGCG

INTERVENTIONS:
Dietary Supplement: green tea extract EGCG — EGCG, 500mg, tid, 4 weeks

SUMMARY:
The aim of this study is to investigate the therapeutic effects of green tea extract on acne treatment and related hormone peptides by a double-blinded, randomized and controlled clinical trial.

DETAILED DESCRIPTION:
change in acne lesions counts, hormone, quality of life

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* 20 to 45 years of age
* moderate or severe acne vulgaris as defined by the Investigator's Global Assessment (IGA; score of 3 or 4 on a scale from 0 to 5)

Exclusion Criteria:

* Received systemic retinoid or hormone treatment in the previous 3 months.
* Abnormal liver enzymes or kidney function tests (1.5 times higher than the upper normal limit)
* abnormal blood chemistry
* Pregnant or breast feeding women or the intention of becoming pregnant
* Concurrent systemic illness
* PCOS
* Very severe acne(IGA score5)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-06 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
acne lesion counts | four weeks

SECONDARY OUTCOMES:
quality of life, SF-12 | four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Hsu CH, Tsai TH, Kao YH, Hwang KC, Tseng TY, Chou P. Effect of green tea extract on obese women: a randomized, double-blind, placebo-controlled clinical trial. Clin Nutr. 2008 Jun;27(3):363-70. doi: 10.1016/j.clnu.2008.03.007. Epub 2008 May 12. PMID 18468736
- [Background] Hsu CH, Liao YL, Lin SC, Tsai TH, Huang CJ, Chou P. Does supplementation with green tea extract improve insulin resistance in obese type 2 diabetics? A randomized, double-blind, and placebo-controlled clinical trial. Altern Med Rev. 2011 Jun;16(2):157-63. PMID 21649457